CLINICAL TRIAL: NCT04911140
Title: Comparison of the Effects of Two Frequencies of Application of Photobiomodulation on Facial Rejuvenation: Controlled, Randomized and Double-Blind Clinical Trial
Brief Title: Comparison of the Effects of Two Frequencies of Application of Photobiomodulation on Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FacialRej
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Wrinkle; Facial Expression
Keywords: photobiomodulation; LED light emitting diode; skin rejuvenation; collagen
MeSH Terms: conditions — Facial Expression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Pre and post treatment assessments will be made by three examiners (three plastic surgeons) who will not be aware of the group in which each patient will be allocated. Participants will not be aware of whether or not they have received the application of the FBM, as they will be using ocular sales. The person responsible for the application will position the equipment in the irradiation locations in all participants and will only activate the light when provided for in the specific experimental group. The characteristic sound of the device will be triggered by recording in the placebos groups for the PBM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Photobiomodulation twice a week (Active Comparator): This group will receive the application of photobiomodulation (PBM) twice a week for 4 weeks.
  Interventions: Radiation: Photobiomodulation twice a week
- Photobiomodulation three times a week (Active Comparator): This group will receive the application of photobiomodulation (PBM) three times a week for 4 weeks.
  Interventions: Radiation: Photobiomodulation three times a week
- Simulated Photobiomodulation (Placebo Comparator): This group will receive the application of simulated photobiomodulation (PBM) twice a week for 4 weeks.
  Interventions: Other: Simulated Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation twice a week — The photobiomodulation will be applied with a LED facial mask, Cosmedical brand (São Paulo, Brazil), containing 92 red LEDs, 660 nm of wavelength, in continuous mode for 21 minutes, twice a week, for 4 weeks.
  Arms: Photobiomodulation twice a week
Radiation: Photobiomodulation three times a week — The photobiomodulation will be applied with a LED facial mask, Cosmedical brand (São Paulo, Brazil), containing 92 red LEDs, 660 nm of wavelength, in continuous mode for 21 minutes, three times a week, for 4 weeks.
  Arms: Photobiomodulation three times a week
Other: Simulated Photobiomodulation — Photobiomodulation will be simulated, with the device turned off, twice a week, for 4 weeks. The characteristic sound of the device will be triggered by recording.
  Arms: Simulated Photobiomodulation

SUMMARY:
Skin aging is an irreversible, slow and progressive process, being influenced mainly by age, but also by external factors such as ultraviolet radiation, smoking, alcohol, among others. Studies have shown benefits of photobiomodulation for facial rejuvenation, especially with the use of red LED. However, there is still a high level of variability in treatment parameters and frequency of application of FBM. The purpose of this study is to compare the effects of photobiomodulation with LED mask (660nm, 6.4 mW/cm², 2.67 J/cm², 5.02 mW, 21 min) on facial rejuvenation using 2 application frequencies: a group will receive 2 weekly applications for 4 weeks and another group will receive 3 weekly applications for the same period. A group with simulated photobiomodulation applied twice a week for 4 weeks will be used as a control. The treatment will be performed in female participants aged between 45 and 60 years. After a period of one month, the depth and width of wrinkles (assessment of face impressions by optical coherence tomography), evaluations of photographic images by specialists (Wrinkle Assessment Scale), as well as the quantitative analysis of the wrinkle size by the Image J software and the level of satisfaction of the participants (FACE-Q) will be compared with data collected before the start of the study. All data will be statistically analyzed according to their distribution, seeking a level of statistical significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers aged 45 to 60 years;
* At menopause (at least 12 months without menstruation);
* Healthy;
* Skin phototype I to IV by Fitzpatrick classification;
* Visible signs of skin aging grades III and IV of the Glogau scale.

Exclusion Criteria:

* With a history of photosensitivity.
* Who have any type of lesion on the skin of the face.
* Who use corticosteroids, anticoagulants, or any drug known to increase photosensitivity, including systemic retinoids and use of topical retinoic acid in the last 6 months.
* People with any collagen-related diseases, malnutrition, anemia, immunosuppression, cancer diseases, smokers, predisposition to hypertrophic and keloid scarring, history of dermatological diseases, surgery on the face, trauma to the face, diseases that could affect the condition of the skin and disease psychiatric.
* Who are in the menstrual period, in the climacteric or in hormone replacement therapy.
* Who underwent cosmetic procedures on the face, such as application of botulinum toxin in the last 8 months, facial filling in the last year, chemical peels, ablative laser and dermabrasion in the last 6 months.
* Who do not respect the post treatment recommendations or who fail to attend a treatment session.
* Those that, during the procedures, present any type of complication (hypersensitivity, allergies) will not be part of the statistical analysis, as these cases will not be in the expected pattern for these procedures. However, these data will be described and discussed, as well as the possible adverse effects and the participants will receive treatment to resolve the condition

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in the scale of evaluation of wrinkles | Baseline and one month after treatment.
  The evaluation of wrinkles will be carried out in a standardized way using the Wrinkle Assessment Scale. In a specific and reserved room, digitalized photographs of the face will be taken in the positions: front, 45 degrees right and left with Canon digital camera model SX510 HS 12.1 MP, using white LED lighting, turquoise blue background, 50cm face distance, manual macro mode, standard that will be followed in the photographs after one month of treatment. The images will be distributed to the three plastic surgeons who will classify them according to the scale of wrinkles and photographic models pre-defined. Each evaluator will receive the same image of wrinkles, all at the end of the experiment. Each image should receive a score from 0 (no wrinkles) to 5 (very deep wrinkles) using the Wrinkle Assessment Scale. The data obtained will be grouped and the evolutionary comparison will be made according to the group of the patient under study.

SECONDARY OUTCOMES:
Changes in wrinkle size (wrinkle width and depth) | Baseline and one month after treatment.
  Before treatment and after 1 month, molds of the frontal lines will be made with light condensation silicone (Clonage, DFL Indústria e Comércio, RJ, Brazil). The silicone mold obtained will be poured into special plaster in a short time. Plaster models will be sent for optical coherence tomography analysis and wrinkle width and depth measured before treatment and after 1 month.
Changes in satisfaction with facial appearance through FACE-Q | Baseline and one month after treatment.
  Participants will answer the FACE-Q questionnaire (satisfaction with facial appearance, adapted for the Portuguese language). FACE-Q is a tool developed to measure the impact and effectiveness of facial aesthetic procedures from the patients' perspective.The results will be tabulated and evaluated according to the sum of the scores obtained in the 10 questions. The higher the score, the more satisfied.
Quantitative evaluation of wrinkles through the measurement of pixels by the Image J software | Baseline and one month after treatment.
  In a specific and reserved room, digitalized photographs of the face will be taken in the positions: front, 45 degrees right and left with Canon digital camera model SX510 HS 12.1 MP, using white LED lighting, turquoise blue background, 50cm face distance and manual macro mode. The quantification in pixels of wrinkles on the forehead, glabellar region, periorbital region and nasolabial fold will be analyzed with Image J software before and after one month of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bragato EF, Paisano AF, Pavani C, Motta LJ, Varellis MLZ, Chiedde M, da Silva GA, Bussadori SK, Mesquita-Ferrari RA, Fernandes KPS. Role of photobiomodulation application frequency in facial rejuvenation: randomized, sham-controlled, double-blind, clinical trial. Lasers Med Sci. 2025 Apr 1;40(1):170. doi: 10.1007/s10103-025-04383-1. PMID 40167796
- [Derived] Bragato EF, Pires JA, Momolli M, Guerra MB, Paisano AF, Ferrari RAM, Bussadori SK, Motta LJ, Fernandes KPS. Comparison of the effects of 2 frequencies of application of photobiomodulation on facial rejuvenation: Controlled, randomized, and double-blind clinical trial. Medicine (Baltimore). 2023 Feb 3;102(5):e32514. doi: 10.1097/MD.0000000000032514. PMID 36749255